CLINICAL TRIAL: NCT03100136
Title: A Non-randomized, Open-label, Exploratory Study With A Non-pharmacologically Active Dose To Evaluate The Binding Kinetics Of A Novel Monoacylglicerol Lipase Positron Emission Tomography Radiotracer [11C]PF-06809247 In Healthy Male Subjects
Brief Title: Test Re-Test Reliability of [11C]PF-06809247 as a Novel PET Tacer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A9001493; PET TRACER METHODOLOGY (Other: Alias Study Number)
Record Dates: First submitted 2017-03-08; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Neuroinflammation
Keywords: PET; [11C]PF-06809247; Reliability; Scan, Safety
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [11C]PF-06809247 (Experimental): A dose intravenous injection of [11C]PF-06809247 followed by PET scanning.
  Interventions: Drug: [11C]PF-06809247

INTERVENTIONS:
Drug: [11C]PF-06809247 — PET Tracer

SUMMARY:
This is a study measuring the binding kinetics and test-retest characteristics of a subpharmacological dose of [11C]PF-06809247 Monoacylglycerol lipase (MAGL) Positron Emission Tomography (PET) tracer in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

-Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease A confirmed positive urine drug test. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.

Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day or 2 chews of tobacco per day.

Screening supine blood pressure greater or equal than140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood. Screening supine 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec.

Subjects with abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary.

Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study treatment. Herbal supplements must be discontinued at least 28 days prior to the first dose of investigational product.

Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.

History of sensitivity to heparin or heparin-induced thrombocytopenia. Unwilling or unable to comply with the Lifestyle Requirements described in the protocol.

Subjects with severe claustrophobia impacting ability to perform the baseline MRI or PET scans.

Fulfillment of any of the MRI contraindications on the standard radiography screening questionnaire (metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos). Any person unable to lie still within the environment of the MRI and PET scanners for the required period to acquire images.

Subjects with any anatomical abnormality in the head that would either preclude or tend to confound the analysis of study data, including any clinically significant abnormal findings from MRI of the head.

Subjects with history of prior radiation exposure for research purposes (eg, x-ray, computer tomography scans, or PET research study(ies)) within the past year Subjects with insufficient arterial patency as determined by Allen's test. Any condition possibly affecting the placement of an intravenous drug administration line, such as poor vein rating as per PCRU procedures. History of sensitivity to local anesthetics likely to be used in the placement of the arterial line.

History of human immunodeficiency virus (HIV), hepatitis B or C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb) and hepatitis C antibody (HCVAb). Male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11-16; Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
binding kinetics of the novel tracer | Day 1, 0, 0:10, 0:20, 0:30, 0:40, 0:50, 1:00, 1:10, 1:20, 1:30, 1:45, 2:00, 2:15, 2:30, 2:45, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 15:00, 20:00, 25:00, 30:00, 45:00, 60:00, 75:00, 90:00, 105:00, 120:00, (min:sec)
  Binding of [11C]PF-06809247 will be assessed by the evaluation of net uptake rate constant Ki (mL/min/g) in the various brain regions modeled, as data permit.

SECONDARY OUTCOMES:
Change in Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 1
  An assessment of Adverse Events
Test - Retest reliability | Day 1
  Test-retest variability of [11C]PF-06809247 binding in the human brain will be assessed using k1, as data permit.
Change in Physical examination | Day 1
  Safety test to check overall health
Change in Neurological Exam | Day 1
  Assessment of sensory neuron and motor responses
Change in 12-lead ECG (electrocardiogram) | Day 1
  heart's electrical activity recorded from electrodes on the body surface
Change in Vital signs | Day 1
  clinical measurements, specifically pulse rate, temperature, and blood pressure, that indicate the state of a patient's essential body functions
Change in Clinical laboratory tests (haematology: haemoglobin; haematocrit/erythrocytes; haemoglobin/erythroctes; Erythro-, leuco-,lympho-, mono-Cytes; Platelets) | Day 1
  Intended to detect, identify, or quantify one or more significant substances, evaluate organ functions, or establish the nature of a condition

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer New Haven Clinical Research Unit, New Haven, Connecticut
  - Anylan Center, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001493&StudyName=A+Non-randomized%2C+Open-label%2C+Exploratory+Study+With+A+Non-pharmacologically+Active+Dose+To+Evaluate+The+Binding+Kinetics+Of+A+Novel+Monoacylglicerol+Lipase+Positron+Emission+Tomography+Radiotracer+%5B11c%5Dpf-06809247+In+Healthy+Male+Subjects